CLINICAL TRIAL: NCT06533774
Title: SpeechSensor and StereoZoom for Pediatrics
Brief Title: Speech Locator_Benefits in Pediatric Popluations
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unreliable data
Sponsor: Sonova AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: eSRF: 7688
Record Dates: First submitted 2024-07-30; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2023-08

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Intervention Model Description: This clinical investigation is an interventional study, executed at one investigation site, with a confirmatory design. The investigation model is single group, with a randomized test order where the test conditions are fully crossed-over.
Masking Description: For objectives 1-3, it is single blinded because all test conditions are implemented in the same hearing aid with the beamformer setting being unknown to the test participant but known to the investigator who enacts program changes.
  For the remaining objectives (4-8), it is non-blinded as participants will be trained on the app before completing a skills test (4), will compare impressions using versus not using the app to change their beamformer (5-7) and speech understanding with versus without amplification (8).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Pediatric Postmarket Surveillance: Yes

ARMS (1):
- Audeo Lumity hearing aid with the SpeechSensor and StereoZoom 2.0 features (Experimental): Audeo Lumity hearing aid and the SpeechSensor and StereoZoom 2.0 features, which is found in the Audeo Lumity devices.
  Interventions: Device: Phonak Audéo Lumity 90-R

INTERVENTIONS:
Device: Phonak Audéo Lumity 90-R — This study will be using the Audeo L90-R devices, which are programmed by the hearing care professional (HCP) using Target fitting software version 8.1.

SUMMARY:
The study seeks to evaluate the impact of SpeechSensor and StereoZoom 2.0 on speech understanding in noise in dynamic listening conditions in pediatric hearing aid users.

DETAILED DESCRIPTION:
The purpose of this study is to substantiate clinical performance claims regarding the benefit of the SpeechSensor feature on speech recognition in noise for side and rear speech as well as StereoZoom 2.0 benefit data for front speech in noise. In addition, the study will yield myPhonak app usability data and claims regarding children's impressions (confidence, anxiety) when given the opportunity to personalize their beamformer settings in noise during a home trial. Finally, this work will confirm hearing aid intended use for pediatric hearing aid users. Results will inform feature setting, provide critical post-market clinical hearing aid data and support for claims.

ELIGIBILITY:
Inclusion Criteria:

* Experienced (> 6 months), full-time hearing aid user
* 10 years up to but not including 18 years of age
* Spoken English
* Ability to understand oral instruction
* Ability to describe listening experiences
* No known neurological issues or cognitive impairment
* Ability to attend the in-person appointment(s)
* No speech/language deficits that could compromising ability to perform tasks
* Healthy outer and middle ear
* Hearing loss consistent with fitting range of the investigational product
* Access to a smartphone that can be used during a home trial
* Informed consent (signature) of parent and consent or assent (verbal) of child

Exclusion Criteria:

* Clinical contraindications (e.g., closed ear canal, absence of pinna)
* Known hypersensitivity or allergy to materials comprising hear-ing aid or acoustic coupling
* Unwilling to wear the hearing aid
* Unwilling or not permitted to use a smartphone
* Aided open-set aided speech recognition scores for speech front (+15 dB SNR) < 30%

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2023-06-08 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Speech intelligibility using AZBio sentences Verbal response accuracy based on percent of words correctly repeated on an open-set sentence recognition in noise task. | 3 hours
  Verbal response accuracy based on percent of words correctly repeated on an open-set sentence recognition in noise task.
  1. Initial - Personalized Signal-to-Noise-Ratio (SNR) is determined for each participant by finding the point where the participant scores 50% correct individual words within sentences. The personalized SNR is determined from the average of two list for a given condition. (SpeechSensor and SZ2.0 objectives)
  2. For comparison conditions - Speech as noise will be presented at the participant's personalized SNR. Speech intelligibility will be determined by accuracy of individual words within sentences. The total words correct is determined for a single list for each condition. (Aided versus unaided, intended use objective).

SECONDARY OUTCOMES:
Speech Focus Slider Usability - Performance on a modified PHAST (Practical Hearing Aid Skills Test) tool will be used to document whether participants can successfully modify the Speech Focus slider. | 3 hours
  1. Ability to use slider in the app will be determined on the basis of successfully or not successfully completing a single task, "In a situation when you want to use the app, show me what you would do." The child will be reinstructed one time and must successfully perform the desired task to be eligible for the home trial.
  2. Ability to successfully use slider in the app will be determined based on successful execution of all of the following tasks correctly):
  i. Show me what you would do to better hear a person in front; ii. Show me what you would do to hear more of the sounds around you. iii. Demonstrate what you should do when you leave the situation.
Preference for having slider | Up to 4 weeks
  Preference for having the Speech Focus slider accessible via the app will be documented with a Yes/ No question on a subjective questionnaire administered post-home trial.
Confidence and Anxiety | Up to 4 weeks
  The possible impact of having access to the Speech Focus slider on confidence and anxiety will be measured using subjective ratings on a post-home trial questionnaire (i.e., Likert scale).

CONTACTS AND LOCATIONS:
Locations (1):
- Hearts for Hearing, Oklahoma City, Oklahoma, United States